CLINICAL TRIAL: NCT03702569
Title: Myocardial Effects of Volume Expansion Evaluated Using Speckle-Tracking (STRAIN) in Intensive Care Unit Patients
Brief Title: Speckle-Tracking and Volume Expansion
Acronym: FLUID-STRAIN
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2018/19
Record Dates: First submitted 2018-10-04; First posted 2018-10-11 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-11

CONDITIONS: Volume Expansion; Left Ventricular Contractility
Keywords: Volume Expansion; Intensive Care Unit; Left Ventricular Contractility; Speckle Tracking; STRAIN
MeSH Terms: conditions — Sprains and Strains

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients needing a volume expansion
  Interventions: Diagnostic Test: Left ventricular global longitudinal strain measure

INTERVENTIONS:
Diagnostic Test: Left ventricular global longitudinal strain measure — Left ventricular global longitudinal strain value measured before and immediately after volume expansion (500mL crystalloid) using speckle tracking images with echocardiography

SUMMARY:
Volume expansion is the cornerstone of hemodynamic management of patients suffering from circulatory failure. The main objective of volume expansion is to increase stroke volume. This increase in stroke volume is due to myocardial contractility improvement. Nowadays, this improvement cannot be assessed using classical monitoring used at the bedside. The main objective of this study is to evaluate left ventricular contractility using Speckle-Tracking before and after volume expansion in intensive care unit patients, to determine if this technology is more sensitive than previous for left ventricular contractility assessment.

DETAILED DESCRIPTION:
The main objective of volume expansion is to increase stroke volume. Frank-Starling curve is schematically divided into two portions: a vertical portion which mean that an increase in preload secondary to volume expansion will induce an increase in stroke volume; and a flat portion which mean that a same increase in preload will not induce an increase in stroke volume. Stroke volume increase is due to a myocardial contractility improvement. Nowadays this improvement cannot be assessed using classical monitoring used at the bedside (left ventricular ejection fraction, fractional area changes, etc …). A new method is available to assess left ventricular contractility at the bedside. Two-dimensional speckle tracking images with echocardiography allows one to track a natural myocardial marker within the myocardium by standard transthoracic echocardiography. It provides unique insights into myocardial function such as tissue deformations and strain rate, which is the rate of deformation. This method is more sensitive than classical echographic left ventricular ejection fraction evaluation. Few data are available about the potential interest of speckle tracking to track an improvement of left ventricular contractility following a volume expansion in intensive care unit patients.

This study is observational, prospective in one center. Patients needing a volume expansion will benefit from an echocardiography (stroke volume and longitudinal strain assessment) before and after fluid challenge (500mL of crystalloids).

The follow up will be restricted to the duration of volume expansion. The last data will be collected just after the end of volume expansion.

ELIGIBILITY:
Inclusion Criteria:

* patient older than 18 years
* hospitalized in neuro-intensive care unit
* volume expansion indicated by the physician
* indication of a transthoracic echocardiography

Exclusion Criteria:

* low echogenicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient older than 18 years hospitalized in neuro-intensive care unit of Bordeaux University Hospital needing volume expansion.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2021-02-17 (Actual); Study Completion 2021-02-17 (Actual)

PRIMARY OUTCOMES:
Left ventricular Global Longitudinal Strain | 3 minutes before the beginning of volume expansion of 500ml of crystalloid
  It is calculated using values of longitudinal strain measured in the three-,four-, and two-chamber of the left ventricle of the heart. GLS is expressed as percentage. Strain is a measure of myocardial muscle fiber shortening during contraction and is calculated as the systolic segment shortening between end-systolic (ES) segment length (L) and end-diastolic (ED) length: strain = (-LES - LED)/LED x 100 %.
Left ventricular Global Longitudinal Strain | 3 minutes after the beginning of volume expansion of 500ml of crystalloid
  It is calculated using values of longitudinal strain measured in the three-,four-, and two-chamber of the left ventricle of the heart. GLS is expressed as percentage. Strain is a measure of myocardial muscle fiber shortening during contraction and is calculated as the systolic segment shortening between end-systolic (ES) segment length (L) and end-diastolic (ED) length: strain = (-LES - LED)/LED x 100 %.
Stroke volume | 3 minutes before the beginning of volume expansion of 500ml of crystalloid
Stroke volume | 3 minutes after the beginning of volume expansion of 500ml of crystalloid

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No